CLINICAL TRIAL: NCT03391427
Title: Ketamine, Lidocaine and Combination for Postoperative Analgesia in Open Liver Resection: A Prospective, Randomized, Four-arm, Double Blind, Placebo Controlled Trial
Brief Title: Ketamine, Lidocaine and Combination for Postoperative Analgesia in Open Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17003
Record Dates: First submitted 2017-12-10; First posted 2018-01-05 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hepatectomy
Keywords: Lidocaine; Ketamine; postoperative analgesia
MeSH Terms: interventions — Lidocaine; Ketamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Lidocaine, ketamine, combination and placebo are being evaluated for treating postoperative pain in major liver resection
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All persons are blinded as the drug is formulated by the investigator who is not the care giver or outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lidocaine (Experimental): This group will receive lidocaine infusion perioperatively
  Interventions: Drug: Lidocaine
- Ketamine (Experimental): This group will receive ketamine infusion perioperatively
  Interventions: Drug: Ketamine
- Lidocaine+ketamine (Experimental): This group will receive a combination of lidocaine and ketamine infusion, perioperatively
  Interventions: Drug: Lidocaine+ketamine
- placebo (Placebo Comparator): This group will receive saline infusion as placebo perioperatively
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — This group will receive lidocaine infusion
  Other Names: Xylocaine; Lidocaine infusion
  Arms: Lidocaine
Drug: Ketamine — This group will receive Ketamine infusion
  Other Names: Ketamine infusion
  Arms: Ketamine
Drug: Lidocaine+ketamine — This group will receive mixture of ketamine and lidocaine infusion
  Other Names: Lidocaine infusion; Ketamine infusion; Xylocaine
  Arms: Lidocaine+ketamine
Drug: Saline — This group will receive saline infusion
  Other Names: Normal saline
  Arms: placebo

SUMMARY:
Lidocaine and ketamine both are being used for perioperative analgesia. Perioperative lidocaine infusion has been shown to reduce postoperative pain and opioid consumption. Perioperative low dose Ketamine has shown improved postoperative pain and reduced opioid usage. We therefore tested the hypothesis that the combination would provide better analgesia in the milieu of intrathecal morphine.

DETAILED DESCRIPTION:
All study participants were monitored according to American Society of Anesthesiologists guidelines. All received intrathecal morphine (300 to 400 mcg) at L3-4 interspace via 25 G Whitacre needle. Participants were then randomized (computer generated) into one of four groups.

General anesthesia was induced and endotracheal intubation was done. Immediately, after intubation, Lidocaine group (L) received a Lidocaine infusion at 0.33 mg/kg/h.

The Ketamine group (K) received a ketamine infusion at 70 mcg/Kg/h. The Lidocaine-Ketamine group (LK) received a Lidocaine infusion at 0.33 mg/kg/h plus a Ketamine infusion at 70 mcg/Kg/h.

The control group (P) received a normal saline infusion to keep the blind. The infusions were stopped approximately 30-45 minute before the completion of surgery.

All participants received a hydromorphone patient-controlled analgesia (PCA) via a pump. All were given acetaminophen 650 mg every 6 hrs for 4 days.

Postoperatively, participants were monitored for nausea, vomiting, sedation, respiratory depression, light-headedness, perioral numbness, pruritus, disturbed dreams and hallucinations.

Postoperative Hydromorphone consumption for the first, second and third day was recorded from the chart maintained by acute pain service team who were blinded to the group assignment.

After the operation, study participants were interviewed at regular intervals by a blinded investigator about their current pain level, as well as satisfaction with pain management. They were also be questioned regarding the presence and severity of opioid-related side effects (nausea, vomiting, sedation, respiratory depression and, pruritus) and light-headedness, perioral numbness, disturbed dreams and hallucinations. Hospital charts were reviewed and data collected to analyze time to request for additional analgesia and total consumption of opioids, non-opioid analgesics, anti-emetics, and antipruritics within the first 72 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 2-4
* Elective major liver resection
* Signed informed consent

Exclusion Criteria:

* ICU admission after surgery
* tracheal extubation not planned after surgery
* language barrier
* mental impairment
* severe coagulopathy
* chronic pain or opioid dependance or both
* alcohol/substance abuse
* allergy to the study drugs
* refusal for spinal
* infection at site of spinal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2015-11-04 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hr
  Total milligrams of opioids consumed would be measured

SECONDARY OUTCOMES:
Opioid consumption | 48 hrs
  Total milligrams of opioids consumed would be measured. Higher opioid consumption indicates worse pain control.
Opioid related side effects | 72 hrs
  Questions regarding all opioid related side effects will be asked. These will include inquiry regarding nausea, vomiting, hallucinations, sedation, respiratory depression, pruritus
Chronic pain | 6 weeks
  Incidence of chronic pain at 6 weeks will be noted by a numerical rating scale of 1-10 where 0 would be no pain at all and 10 would be worst possible pain. This is standard pain assessment tool. Lower numbers indication better outcomes.
Patient satisfaction | 72 hrs
  Patient satisfaction will be noted using a numeric rating scale; where 0 will be completely unsatisfied and 10 will be completely satisfied. Higher values depict better satisfaction and better outcomes.
Chronic pain | 12 weeks
  Incidence of chronic pain at 12 weeks will be noted by a numerical rating scale of 1-10 where 0 would be no pain at all and 10 would be worst possible pain. This is standard pain assessment tool. Lower numbers indication better outcomes.
Opioid consumption | 72 hrs
  Total milligrams of opioids consumed would be measured. Higher opioid consumption indicates worse pain control.

CONTACTS AND LOCATIONS:
Overall Officials: Achal Dhir, Principal Investigator — Lawson
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Background] Harvey KP, Adair JD, Isho M, Robinson R. Can intravenous lidocaine decrease postsurgical ileus and shorten hospital stay in elective bowel surgery? A pilot study and literature review. Am J Surg. 2009 Aug;198(2):231-6. doi: 10.1016/j.amjsurg.2008.10.015. Epub 2009 Mar 12. PMID 19285304
- [Background] Rakic AM, Golembiewski J. Low-dose ketamine infusion for postoperative pain management. J Perianesth Nurs. 2009 Aug;24(4):254-7. doi: 10.1016/j.jopan.2009.05.097. No abstract available. PMID 19647665
- [Background] Ko JS, Choi SJ, Gwak MS, Kim GS, Ahn HJ, Kim JA, Hahm TS, Cho HS, Kim KM, Joh JW. Intrathecal morphine combined with intravenous patient-controlled analgesia is an effective and safe method for immediate postoperative pain control in live liver donors. Liver Transpl. 2009 Apr;15(4):381-9. doi: 10.1002/lt.21625. PMID 19326422